CLINICAL TRIAL: NCT02913079
Title: The Acute Impact of Sit-stand Desks on Post-meal Blood Sugar Levels
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Prince Edward Island (Other)
Responsible Party: Principal Investigator, Travis Saunders, Assistant Professor, University of Prince Edward Island
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 6006774
Record Dates: First submitted 2016-09-15; First posted 2016-09-23 (Estimated); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Insulin Sensitivity; Glucose Tolerance; Sedentary Behaviour; Physical Activity
MeSH Terms: conditions — Insulin Resistance; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sit-stand desk (Experimental): During this condition, participants will sit or stand as much as they like throughout a workday.
  Interventions: Behavioral: Sit-stand desk
- Sitting (Placebo Comparator): During this condition, participants will work in the sitting position only.
  Interventions: Behavioral: Sitting desk

INTERVENTIONS:
Behavioral: Sit-stand desk
  Arms: Sit-stand desk
Behavioral: Sitting desk
  Arms: Sitting

SUMMARY:
Context and Rationale: Uninterrupted sitting is associated with increased risk of diabetes, heart disease, and death, even among people who are physically active. These relationships are likely due to increases in post-meal blood sugar observed when people sit for long periods (e.g. > 1 hour) without interruption. In contrast to sitting, standing results in large reductions in post-meal blood sugar levels. Our group has recently shown that sit-stand desks result in large (e.g. 2.5 hour/day) reductions in occupational sitting time. Taken together, these findings suggest that sit-stand desks may help to reduce post-meal blood sugar levels. However, this has yet to be examined in the field. Theoretical Approach and Objectives: The objective of this randomized crossover study is to determine whether people have lower blood sugar when using a sit-stand desk, in comparison to a desk that can only be used while sitting. Methods and Procedures: Sixteen participants will be asked to wear a continuous glucose monitor to measure their blood sugar levels during 2 separate conditions. During one condition, they will be asked to use a sit-stand desk to sit and/or stand as much as they like during 1 workday. During the other condition, they will be asked to work at a seated desk for 1 workday. Participants will be provided with identical meals to eat during each of the two conditions. We hypothesize that participants will have lower blood sugar levels on the day when they use the sit-stand desk, in comparison to the day using a traditional seated desk. Significance and Future Use: If our results support this hypothesis, this would suggest that sit-stand desks may be a useful way to reduce blood sugar levels in people at risk for diabetes. This could also lead to larger population-based interventions studying the health impact of sit-stand desks.

ELIGIBILITY:
Inclusion Criteria:

* To participate in this study, participants must be between the ages of 20 and 65, and have access to a sit-stand desk (depending on your workspace, we may be able to provide you with a sit-stand desk during the study if you do not already have one).

Exclusion Criteria:

* Participants will be excluded if they are currently taking any diabetes medications targeting blood sugar or insulin sensitivity as this will impact our primary outcome of postprandial glucose. Participants will also be excluded if they are unable to stand or walk independently, as these are secondary outcomes in the present study.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2016-09; Primary Completion 2018-06 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Postprandial Glucose | 12 hours
  Postprandial glucose will be assessed over 1 workday in both the experimental and control conditions.

SECONDARY OUTCOMES:
Objectively measured minutes of light, moderate and vigorous physical activity. | 24 hours
  Physical activity time will be assessed over 1 workday during both conditions.
Objectively measured minutes of sitting | 24 hours
  Sitting time will be assessed over 1 workday during both conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Prince Edward Island, Charlottetown, Prince Edward Island, Canada

IPD SHARING:
Plan to Share IPD: No
No.